CLINICAL TRIAL: NCT03142633
Title: MicroRNA as Biomarkers for Development of Metabolic Syndrome in Women With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-525
Record Dates: First submitted 2017-03-20; First posted 2017-05-05 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Buffy Coat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Polycystic Ovary Syndrome: Participants of the PICOLO study
  Inclusion criteria:
  Women aged 18-40 years when included in the PICOLO-cohort, PCOS based on the Rotterdam 2003 consensus criteria Exclusion criteria: Contraceptive pills within 6 weeks from examination, endocrinological disease (i.e. diabetes, thyroid dysfunction), endometriosis and premature ovarian insufficiency, breastfeeding women and pregnancy.

SUMMARY:
The aim of this study is to explore the microRNA profile in serum of women with Polycystic Ovary Syndrome and investigate the correlation between the microRNA profile and markers of metabolic syndrome.

DETAILED DESCRIPTION:
The study consist of 2 parts:

1. A cross-sectional study of a cohort of women with PCOS with analysis of materials from the established biobank. (the PICOLO cohort) Data and blood samples from 266 women with PCOS was collected from January 2010 - February 2013 as a part of the PICOLO collaboration: "PCOS, infertility, Cardiovascular and Obstetric risk markers and Long-term Outcome" at Holbaek Fertility Clinic and at Herlev Hospital.

   Serum samples will be analysed with Reverse Transcript polymerase chain Reaction (RT-qPCR) for selected microRNAs.
2. A follow-up study of local participants from the PICOLO study. 90 of the participants were recruited at Holbaek Fertility Clinic.

Following tests will be performed at reexamination, in order to describe the clinical phenotype: Health interview, anthropometrics, acne score, Ferriman-Gallway score, blood pressure, Transvaginal ultrasound of uterus and ovaries, insulin Resistance (IR) assessed with Oral glucose Tolerance test (OGTT), Venous blood for hormone analysis and lipid status.

MicroRNA analysis with Taqman microRNA array will be performed on serum samples.

Detection and treatment of women with PCOS is a challenge due to the variability of the syndrome. If MiRNA could serve as marker of metabolic syndrome, it would be possible to detect and follow the women of greater risk at an earlier stage, and thereby preventing morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years when included in the PICOLO study
* PCOS based on the Rotterdam 2003 consensus criteria

Exclusion Criteria:

* Contraceptive pills within 8 weeks from examination,
* endocrinological disease (i.e. type 1 diabetes thyroid dysfunction),
* Severe endometriosis (stage III and IV)
* Premature ovarian insufficiency,
* Breastfeeding women and
* Pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Local Participants from the PICOLO study, performed at Holbæk Hospital between 2010 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
MicroRNA profile | MicroRNA analysis will be performed on serum from baseline visit (biobank material) and on serum obtained from a follow-up visit 5 years after baseline. The participants will be examined for 2 hours at follow up.
  The change in relative expression of MicroRNA in women with PCOS will be assessed, using TaqMan microRNA arrays, comparing serum samples from baseline from an existing biobank with serum samples from a follow up visit.

SECONDARY OUTCOMES:
Insulin Resistance and Type 2 Diabetes | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Insulin Resistance will be assessed by Oral glucose Tolerance test (OGTT). Venous blood samples and measurement of glucose, serum insulin and C-peptid will be collected at -5, 0, 30 and 120 min after a 75 g glucose load. Impaired glucose tolerance will be assessed by calculation of BIGTTs1(insulin sensitivity index) and BIGTTAIR(Acute insulin response)
Blood Pressure | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Evaluated > 140/90 mmHg
Abdominal obesity | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Waist-Hip Ratio. Elevated > 0,85
Overweight | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Defined: BMI > 25 kg/m2
Dyslipidemia | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Defined as triglycerides > 1,7mmol/L, Total cholesterol > 5,0, LDL > 3,0 or HDL<1,0 mmol/L
PCOS status | The participants will be examined for 2 hours, at a follow-up visit 5 years after the baseline visit.
  Evaluated by Rotterdam (2003) criteria:
  1. Polycystic Ovaries:Number of antral follicles >12, ovarian volume (length*depth*width/2) > 10 mL 2) Clinical (evaluated by Ferriman Gallway score) or biochemical signs of hyperandrogenism ( Free Testosterone > 0.034 nmol/Lor total testosterone >1.8 nmol/L) 3.Oligo or amenorrhea ´(>35 days between bleedings)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lis M Englund, DsMC, Principal Investigator — Fertility Clinic, Dept. of Gynecology and Obstetrics, Holbæk Hospital
Locations (1):
- Fertility Clinic,Department of Gynecology and Obstetrics, Holbæk, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Udesen PB, Sorensen AE, Svendsen R, Frisk NLS, Hess AL, Aziz M, Wissing MLM, Englund ALM, Dalgaard LT. Circulating miRNAs in Women with Polycystic Ovary Syndrome: A Longitudinal Cohort Study. Cells. 2023 Mar 23;12(7):983. doi: 10.3390/cells12070983. PMID 37048055
- [Derived] Udesen PB, Sorensen AE, Joglekar MV, Hardikar AA, Wissing MLM, Englund AM, Dalgaard LT. Levels of circulating insulin cell-free DNA in women with polycystic ovary syndrome - a longitudinal cohort study. Reprod Biol Endocrinol. 2019 Apr 5;17(1):34. doi: 10.1186/s12958-019-0478-7. PMID 30953560